CLINICAL TRIAL: NCT02208297
Title: Study to Assess Loteprednol Etabonate Ophthalmic Gel, 0.38% Versus Vehicle Gel for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery
Brief Title: Loteprednol Etabonate Ophthalmic Gel for the Treatment of Ocular Inflammation and Pain Following Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 843
Record Dates: First submitted 2014-08-01; First posted 2014-08-05 (Estimated); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Inflammation; Pain; Cataract
MeSH Terms: conditions — Inflammation; Pain; Cataract | interventions — BID protein, human; Loteprednol Etabonate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol Etabonate Gel (BID) (Experimental): Loteprednol Etabonate Gel 0.38% administered two times daily (BID)
  Interventions: Drug: Loteprednol Etabonate Gel (BID)
- Vehicle Gel (BID) (Placebo Comparator): Vehicle gel administered two times daily (BID)
  Interventions: Drug: Vehicle Gel (BID)

INTERVENTIONS:
Drug: Loteprednol Etabonate Gel (BID) — One drop of LE gel instilled into the study eye two times per day (BID) for 14 days
  Other Names: Lotemax
  Arms: Loteprednol Etabonate Gel (BID)
Drug: Vehicle Gel (BID) — One drop of vehicle gel instilled into the study eye two times per day (BID) for 14 days
  Other Names: Vehicle
  Arms: Vehicle Gel (BID)

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of loteprednol etabonate (LE) ophthalmic gel, 0.38% (BID)

DETAILED DESCRIPTION:
The objective of this study is to evaluate the safety and efficacy of loteprednol etabonate (LE) ophthalmic gel, 0.38% (BID) for the treatment of inflammation and pain following cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

Visit 1 (Screening Visit)

* Be willing and able to comply with all treatment and follow-up/study procedures.
* Be a candidate for routine, uncomplicated cataract surgery.

Visit 3 (Postoperative Day 1)

* Have undergone routine, uncomplicated cataract surgery (phaco-emulsification with posterior chamber intraocular lens (IOL) implantation, not combined with any other surgery) in the study eye.
* Have ≥ Grade 2 anterior chamber (AC) cells (6-15 cells) in the study eye.

Exclusion Criteria:

* Have a severe/serious ocular condition or history/presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the result(s) of the study.
* Have known hypersensitivity or contraindication to the study drug(s) or their components.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2014-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Vittitow, Study Director — Valeant/Bausch & Lomb
Locations (1):
- Bausch & Lomb Incorporated, Bridgewater, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Loteprednol Etabonate Gel (BID) | Vehicle Gel (BID)
Started | 163 | 163
Completed | 141 | 107
Not Completed | 22 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Loteprednol Etabonate Gel (BID) | Vehicle Gel (BID) | Total
Number analyzed (Participants) | 163 | 163 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (9.88) | 67.8 (8.45) | 67.4 (9.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 101 | 190
  Male | 74 | 62 | 136

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells
Description: White blood cell accumulation in anterior aqueous humor was assessed by the Investigator during slit lamp examination and graded on a 5-point scale: Grade 0 = no cells seen; Grade 1 = 1 to 5 cells; Grade 2 = 6 to 15 cells; Grade 3 = 16 to 30 cells; Grade 4 = > 30 cells. Lower score indicated better outcome. Complete resolution of AC cells was defined as cell score = 0 in the study eye.
Time Frame: 8 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Loteprednol Etabonate Gel (BID) | Vehicle Gel (BID)
Number analyzed (Participants) | 163 | 163
Participants | 38 | 29

2. Primary Outcome: Percentage of Participants With Grade 0 Pain in the Study Eye.
Description: Ocular pain, defined as a positive sensation of the eye, including foreign body sensation, stabbing, throbbing, or aching, was assessed and graded by subjects on the 6-point scale, with 0=None and 5=Severe.
Time Frame: 8 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Loteprednol Etabonate Gel (BID) | Vehicle Gel (BID)
Number analyzed (Participants) | 163 | 163
Participants | 120 | 97

3. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells by Visit
Description: as for outcome 1
Time Frame: 18 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Loteprednol Etabonate Gel (BID) | Vehicle Gel (BID)
Number analyzed (Participants) | 163 | 163
Participants
  Day 3 | 16 | 11
  Day 15 | 82 | 57
  Day 18 | 80 | 67

4. Secondary Outcome: Percentage of Participants With Grade 0 Pain in the Study Eye by Visit.
Description: as for outcome 1
Time Frame: 18 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Loteprednol Etabonate Gel (BID) | Vehicle Gel (BID)
Number analyzed (Participants) | 163 | 163
Participants
  Day 8 | 106 | 87
  Day 15 | 132 | 95
  Day 18 | 122 | 91

5. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Flare in the Study Eye by Visit.
Description: Flare was evaluated by the Investigator by assessing the scattering of a slit lamp light beam directed into the anterior chamber (Tyndall effect). Flare was graded on the 5-point scale, with 0=None (best) and 4=Very Severe (worst). Complete resolution of AC flare was defined as Grade 0.
Time Frame: 18 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Loteprednol Etabonate Gel (BID) | Vehicle Gel (BID)
Number analyzed (Participants) | 163 | 163
Participants
  Day 1 | 96 | 71
  Day 8 | 114 | 81
  Day 15 | 131 | 100
  Day 18 | 128 | 98

6. Secondary Outcome: Percentage of Participants With Complete Resolution of Anterior Chamber (AC) Cells and AC Flare in the Study Eye by Visit.
Description: White blood cell accumulation in anterior aqueous humor was assessed by the Investigator during slit lamp examination and graded on a 5-point scale: Grade 0 = no cells seen; Grade 1 = 1 to 5 cells; Grade 2 = 6 to 15 cells; Grade 3 = 16 to 30 cells; Grade 4 = > 30 cells. Lower score indicated better outcome. Complete resolution of AC cells was defined as cell score = 0 in the study eye. Flare was evaluated by the Investigator by assessing the scattering of a slit lamp light beam directed into the anterior chamber (Tyndall effect). Flare was graded on the 5-point scale, with 0=None (best) and 4=Very Severe (worst).
Time Frame: 18 days
Population: The analysis population included all randomized participants, with missing values imputed as non-responders.
Measure: Count of Participants; unit: Participants
Arm/Group | Loteprednol Etabonate Gel (BID) | Vehicle Gel (BID)
Number analyzed (Participants) | 163 | 163
Participants
  Day 3 | 15 | 9
  Day 8 | 37 | 29
  Day 15 | 80 | 56
  Day 18 | 80 | 67

ADVERSE EVENTS:
Time Frame: 18 days
Description: The safety analysis population included all randomized participants who received treatment. There was one participant who did not receive treatment, thus there were 325 participants in the safety population.
Arm/Group | Loteprednol Etabonate Gel (BID) | Vehicle Gel (BID)
All-Cause Mortality (participants affected / at risk) | 0/162 | 0/163
Serious Adverse Events (participants affected / at risk) | 0/162 | 1/163
Other Adverse Events (participants affected / at risk) | 0/162 | 0/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Loteprednol Etabonate Gel (BID) (N=162) | Vehicle Gel (BID) (N=163)
Endophthalmitis (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.